CLINICAL TRIAL: NCT05044936
Title: The Effects of Topical Cannabidiol Cream on Post-exercise Recovery
Brief Title: Topical Cannabidiol Cream and Post-exercise Recovery
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The researchers were not able to acquire funding to initiate the study. Also, the study was not approved by the local IRB which requested a FDA new drug application.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBD2021
Record Dates: First submitted 2021-07-21; First posted 2021-09-16 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Muscle Damage
Keywords: Exercise; Resistance training; Canabidiol
MeSH Terms: conditions — Motor Activity | interventions — Cannabidiol; Resistance Training; Exercise

STUDY DESIGN:
Intervention Model Description: Repeated Measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Training (Experimental): Visit 1: sign consent form, pregnancy tests for females, resting blood pressure, height/weight, body composition, and VO2max test. Visit 2: 1-repetition maximum (RM) test and protocol familiarization. Visit 3: perform a muscle-damaging exercise protocol. Pre-exercise soreness and blood samples will be collected. After, they will perform the pre-exercise testing to assess baselines levels of power and sprint times. Upon completion, they will undergo the muscle-damaging exercise protocol. Post-exercise blood samples and soreness will be collected. The participant will then be given either placebo or CBD cream to rub into their quadriceps. Visit 4 & 5: collect blood samples and soreness scale measurements. Participants will then be given the same treatment (placebo or CBD cream) as they had on visit 3. Visit 6 will be similar to visit 3, except the participant will be given the opposite treatment (placebo or CBD cream). Visits 7 & 8 will be similar to visits 4 & 5, respectively.
  Interventions: Drug: Cannabidiol Oil; Other: Resistance Exercise

INTERVENTIONS:
Drug: Cannabidiol Oil — The dose that will be used for each administration of CBD will be 0.5mg/kg of body mass. As there are no recommendations for CBD from the FDA or through previous research in humans, and especially for CBD cream, the dosage is based on the United Kingdom's governing body recommending maximal amounts of CBD ingestion being 1 mg/kg per day. Further, the "practical" amount that companies "recommend" is anywhere from a "pea size" to a "handful," which can range from high and low amounts. Using 0.5mg/kg of body mass allows for a moderate use of the lotion, as well as leaving extra quantities throughout the day should people want to use CBD outside of their post-workout recovery strategies outside of a laboratory setting. To convert the amount of CBD to the amount of lotion, we will divide the amount of CBD (0.5 mg/kg) by 4.85 (the amount of mg of CBD per gram of lotion). This will calculate the amount (in grams) of lotion each participant will receive.
  Other Names: CBD
Other: Resistance Exercise — Participants will complete eccentric-based leg press (4-s lowering phase and 1-s upward phase) for 10 sets of 8 repetitions at 70% 1RM in order to induce muscle damage using a leg press machine. Three minutes of rest will be permitted between sets. Following the 10th leg press, participants will complete 4 sets of 20 consecutive plyometric lunges using only their body weight. Two minutes of rest will be permitted between sets. The muscle damaging protocol will be done upon completion of the 4th set of plyometric lunges.
  Other Names: Exercise

SUMMARY:
This proposal's objective is to investigate the effects of topical cannabidiol (CBD) cream on exercise-induced muscle damage, exercise-induced inflammatory markers, and subsequent exercise performance after an exercise-induced damage protocol.

DETAILED DESCRIPTION:
Intro Canabidiol (CBD), a non-intoxicating cannabinoid, has recently stimulated great interest in the scientific community with an increased number of publication in the last decade. While it was first isolated and reported in 1963, subsequent studies were not published until the late 2000s. These studies have mainly focused on the effects of CBD on pain management, and anti-inflammatory processes Current evidence indicates that CBD plays a role in anti-inflammatory and antioxidant processes. CBD has been shown to act as an agonist for ionotropic cannabinoid receptors including chemo- and thermosensitive members of the Transient Receptor Potential (TRP) channel superfamily. This is important as this mechanism may decrease neuropeptide expression, and in turn decreases the release of pro-inflammatory cytokines and chemokines such as interleukin 1 alpha (IL-Iα), interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-α), and cyclooxygenase-2 (COX-2).

The application of CBD use varies, as it can be consumed orally as an oil, inhaled as a high concentration vape oil, or be applied topically. Although oral bioavailability of CBD is limited, recent research has shown that a single, oral dose (1500-6000mg) can still reach peak plasma concentrations of ~0.9 - 2.5 micrometers (uM) within ~4-5 hours with a half-life of ~14-17 hours (Taylor et al., 2018). Further, evidence suggests that ingested CBD can have a significant influence on the delayed onset of muscle soreness due to exercise-induced muscle damage, though the exact mechanisms were not. Conversely, recent evidence suggests that 150 mg of CBD oil had no effect on non-invasive markers of muscle damage in untrained men after 24 and 48 hours post-exercise. While inhaled CBD has not been studied thoroughly, a recent study in which participants vaporized 100 mg of CBD observed high blood CBD concentrations (104.6 ng/mL) after 30 minutes, although terminal half-life and max concentrations were not collected (Spindle et al., 2020). Still, an insufficiency in data regarding inhaled CBD is apparent. Given the low bioavailability of oral ingestion of CBD and the lack of research in inhaled CBD, the transdermal application may be an effective option. CBD has successfully been delivered transdermally in different animal species for anti-inflammatory activity and has indicated that topical application of CBD gel is an effective treatment for reduction in inflammation and hypersensitivity in rats. Specifically, research showed that a 6.2 mg/day dose optimally reduced swelling, while higher values (62.3 mg/day) did not yield additional improvements. These studies demonstrate transdermal administration of CBD may have therapeutic effects, although more research is necessary, especially as it pertains to humans.

In the context of sports, CBD's recent removal from the Prohibited List of the World Anti-Doping Agency (WADA) has no doubt aided in the increased use of CBD, especially considering that CBD is safe and well-tolerated at high doses (1,500 mg/day) or as an acute dose of 6,000mg. However, there are currently little evidence indicating that CBD may exert an ergogenic effect or accelerate/facilitate muscle recovery. In regard to potential ergogenic effects, no studies exist. While CBD may play a role in glucose metabolism and lipid storage via activation of Peroxisome proliferator-activated receptor ( PPARy), as well as increased activity of mitochondrial complexes, no data exists stating that it would aid in performance as an ergogenic. Thus, the majority of CBD use and studies have focused on recovery.

While CBD has been reported to exert a number of physiological, biomechanical, and psychological effects, the specific effects on human skeletal muscle, exercise recovery, and subsequent exercise performance are limited. Cannabinoid receptors (CB1) activation has been shown to increase AMP-activated kinase a1 (AMPKa1) messenger ribonucleic acid (mRNA) expression, which suggests that CB1 receptors are active in skeletal muscle. Still, these data are inconsistent, as blocking of CB1 pathways plays a permissive role for Anandamide (AEA) stimulation of AMP-activated kinase a2 (AMPKa2) in lean subjects, but it plays an inhibitory role in obese subjects.

In regard to exercise recovery, there is evidence in animal and cell studies that CBD may limit the harmful effects of inflammation by decreasing immune cell accumulation, stimulating production of anti-inflammatory cytokines, inhibiting production of pro-inflammatory cytokines, and attenuating reactive oxygen species. There is also evidence that CBD acts directly on muscle plasticity affecting quality and performance by modulating levels of myogenin and troponin-t-1 transcription levels. Further, evidence suggests CBD causes a significant reduction in all myogenic transcripts but does not reduce the expression of muscle differentiation markers, which may suggest it can attenuate inflammation without blunting muscular adaptations. In regard to the use of CBD on post-exercise markers in humans, there is evidence suggesting that the use of CBD can decrease delayed-onset muscle soreness (DOMS), although an apparent paucity exists. Comparatively, other evidence suggests that the use of CBD has no effect on DOMS, especially in untrained males. Exercise, especially when strenuous, and with a heavy eccentric component, can cause acute damage to skeletal muscle myofibrils and the surrounding extracellular matrix. Exercise-induced muscle damage (EIMD) can impair muscle function and initiate an inflammatory response. Although inflammation is necessary for EIMD repair and adaptation, excessive inflammation attenuates functional recovery and may contribute to prolonged muscle soreness. Based on the evidence from cell and animal studies, CBD could reduce inflammation and facilitate muscle recovery.

Although recent developments in the effects of CBD on modulation of inflammatory processes have occurred, there remains a paucity in its specific use for exercise. It is suggested that the availability of transdermal CBD, as well as the ease of its applicability, makes it the logical next step in research. Further, transdermal delivery of CBD has been investigated, but not within the context of exercise performance and EIMD. Therefore, the purpose of this study will be to assess the efficacy of transdermal application of CBD delivery to reduce pain-related behaviors and decrements in exercise performance associated with EIMD. It is hypothesized that transdermal application of CBD will decrease pro-inflammatory and increase blood anti-inflammatory markers, and attenuate decrements in subsequent exercise performance after an exercise-induced damage protocol.

Methods Experimental Approach Utilizing a randomized, double-blind experimental design, participants will be assigned to using transdermal application of a cream with either 1 g of CBD or placebo upon completion of exercise. Muscle soreness, venous blood (for the assessment of creatine kinase (CK) and lactate dehydrogenase (LDH) will be collected prior to eccentric exercise, immediately post, and 1-, 4-, 24-, and 48-h post-exercise. After 48 hours, muscle function will be assessed by general sports testing.

Subjects Subjects will be 24 apparently healthy, resistance-trained, and aerobically fit males and females. All subjects will self-report via Healthy History questionnaire and Physical Activity Readiness Questionnaire (PARQ) that they participate in >150 weekly minutes of moderate-to-vigorous exercise, which included a blend of aerobic and resistance training. Subjects will report that they are free of cardiovascular, metabolic, viral, kidney, and liver disease with no orthopedic injuries that would prevent them from exercise. Furthermore, subjects will need to have engaged in at least two days/week of total-body resistance exercise for > 6 months. All subjects will self-report that they are familiar with the resistance exercise (RE) performed in this study and they have had previous experience with eccentric training. Before experimental trials begin, height (cm) and body mass (kg) will be measured without shoes using a stadiometer to the nearest 1 cm, and a scale to the nearest 0.1kg, respectively. Additionally, body fat percentage (BF%) will be measured using a 3-site skinfold: chest, abdomen, and thigh for males and triceps, suprailiac, and thigh for females. These values will be used to estimate body density and BF%.

Procedures

1 Repetition Maximum (1RM) Determination Before performing each exercise, proper lifting technique and cadence will be demonstrated by a researcher who is certified by the National Strength and Conditioning Association (NSCA), American College of Sports Medicine (ACSM), or National Athletic Training Association. After observing proper form and descriptions of each exercise, subjects will perform 5-10 minutes of a self-selected warm-up before executing the first set of RE with ~50% of their self-estimated 1RM for 8-10 repetitions. Following a 3-5 min rest period, successive sets will be performed, and researchers will continue to add weight for each set until a successful 1RM is determined. A rest period of 3-5 minutes will be provided between each set, as recommended by the NSCA. All 1RM's will be determined within three attempts, within the same day. The 1RM will be determined for the leg. Subjects will be given 3-5 minutes of rest between exercises.

Resistance Exercise Protocol Participants will complete eccentric-based leg press (4-s lowering phase and 1-s upward phase) for 10 sets of 8 repetitions at 70% 1RM in order to induce muscle damage using a leg press machine. Three minutes of rest will be permitted between sets. Following the 10th leg press, participants will complete 4 sets of 20 consecutive plyometric lunges using only their body weight. Two minutes of rest will be permitted between sets. The muscle damaging protocol will be done upon completion of the 4th set of plyometric lunges.

Muscle-Damaging Exercise Visit Upon arrival to the laboratory, pre-exercise blood samples will be collected. Pre-exercise perceived soreness, vertical jump, maximum voluntary contraction (MVC), maximum voluntary isometric contraction (MVIC), and 10-yard sprint will be tested. Participants will then complete a 10-min self-selected dynamic warm-up followed by the muscle-damaging squat exercise protocol. Following completion of the exercise protocol, participants will have their blood drawn, and their rating of perceived muscle soreness taken.

Blood Collection, Perceived Soreness, and Muscle Performance Blood Collection and Assessments Blood will be collected pre-muscle damaging exercise, post-exercise, 1-, 4-, 24-, and 48-H post-exercise for the collection of plasma. Blood samples will be collected from the antecubital vein, centrifuged at 1650x g for 10 min, and stored at -80 C until analysis. As indirect markers of muscle damage, plasma concentrations of CK and LDH will be determined at pre-muscle-damaging exercise, 4-, 24-, and 48-H. CK and LDH will be determined in duplicate using enzymatic assays according to the manufacturer's guidelines.

Perceived Soreness A paper-version visual analog scale will be used to assess perceived soreness. Zero centimeters will represent no soreness, while 10 cm will represent extreme soreness. Participants will rate their perceived soreness at all time points (pre-exercise, post-exercise, 1-, 4-, 24-, and 48-H).

MVC Using the Biodex System, participant's MVC strength of the dominant limb knee extensor will be assessed. Each participant's Biodex chair position will be kept standard for all visits and attempts. The participant's knee will be placed at 120° of flexion. Three 5-s contractions will be completed with one minute of rest between attempts. The attempt resulting in the highest peak torque (newton-meters) will be recorded and used for statistical analysis.

Maximal Voluntary Isometric Contraction Using the Biodex System, participant's MVIC strength of the dominant limb knee extensor will be assessed. Each participant's Biodex chair position will be kept standard for all visits and attempts. The participant's knee will be placed at 120° of flexion. Three 5-s contractions will be completed with one minute of rest between attempts. The attempt resulting in the highest peak torque (newton-meters) will be recorded and used for statistical analysis.

Vertical Jump Vertical jump will be assessed using a Tendo Unit (Tendo Sport; London, UK.) by attaching it to the participant and instructing them to jump. Participants will be allowed three jumps, with the jump with the highest power output, recorded used for statistical analysis. Two minutes of rest will be given between attempts.

Ten-yard sprint Participants will be asked to sprint 10 yards as fast as possible in a straight line. They will be instructed to begin with their preferred foot forward and placed on a line taped on the floor from a standing position. The same forward foot will be used for all test time points. Participants will perform three sprints and an automatic digital timer linked to sensors (Bower Timing Systems, Draper, UT) will be placed at the 0- and 10yd marks to assess the total sprint time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, recreationally trained young adult-aged females and males
* Been engaging in resistance training (> 2 days/weeks for > 6 months)
* Classified as "low risk" according to criteria put forth by American College of Sports Medicine

Exclusion Criteria:

* Cardiovascular, metabolic, viral, kidney, liver disease, or acute orthopedic injuries
* Pregnant or planning to become pregnant during the study
* Unable to consent
* Under 18 years of age
* Over 35 years of age
* Prisoners
* Participants with cognitive impairment or with legally authorized representative

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in indirect markers of muscle damage | 24 & 48 hours post-training
  Measuring lactate dehydrogenase blood levels
Change in indirect markers of muscle damage | 24 & 48 hours post-training
  Measuring creatine kinase blood levels
Change in muscle soreness | 24 & 48 hours post-training
  Measuring using a soreness visual analog scale from 0-10, where 0 means no soreness, and 10 means extremely high/painful levels of soreness
Change in exercise performance | 24 & 48 hours post-training
  Measure differences in maximum voluntary contraction.
Change in exercise performance | 24 & 48 hours post-training
  Measure differences in vertical jump
Change in exercise performance | 24 & 48 hours post-training
  Measure differences in sprint time

CONTACTS AND LOCATIONS:
Overall Officials: Fabiano Amorim, PhD, Study Chair — University of New Meixoco
Locations (1):
- UNM Exercise Physiology Lab, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonn-Miller MO, Loflin MJE, Thomas BF, Marcu JP, Hyke T, Vandrey R. Labeling Accuracy of Cannabidiol Extracts Sold Online. JAMA. 2017 Nov 7;318(17):1708-1709. doi: 10.1001/jama.2017.11909. PMID 29114823
- [Background] Burstein S. Cannabidiol (CBD) and its analogs: a review of their effects on inflammation. Bioorg Med Chem. 2015 Apr 1;23(7):1377-85. doi: 10.1016/j.bmc.2015.01.059. Epub 2015 Feb 7. PMID 25703248
- [Background] Cavuoto P, McAinch AJ, Hatzinikolas G, Cameron-Smith D, Wittert GA. Effects of cannabinoid receptors on skeletal muscle oxidative pathways. Mol Cell Endocrinol. 2007 Mar 15;267(1-2):63-9. doi: 10.1016/j.mce.2006.12.038. Epub 2006 Dec 21. PMID 17270342
- [Background] Clarkson PM, Nosaka K, Braun B. Muscle function after exercise-induced muscle damage and rapid adaptation. Med Sci Sports Exerc. 1992 May;24(5):512-20. PMID 1569847
- [Background] Cochrane-Snyman KC, Cruz C, Morales J, Coles M. The Effects of Cannabidiol Oil on Noninvasive Measures of Muscle Damage in Men. Med Sci Sports Exerc. 2021 Jul 1;53(7):1460-1472. doi: 10.1249/MSS.0000000000002606. PMID 33481484
- [Background] Fatouros IG, Jamurtas AZ. Insights into the molecular etiology of exercise-induced inflammation: opportunities for optimizing performance. J Inflamm Res. 2016 Oct 21;9:175-186. doi: 10.2147/JIR.S114635. eCollection 2016. PMID 27799809
- [Background] Hammell DC, Zhang LP, Ma F, Abshire SM, McIlwrath SL, Stinchcomb AL, Westlund KN. Transdermal cannabidiol reduces inflammation and pain-related behaviours in a rat model of arthritis. Eur J Pain. 2016 Jul;20(6):936-48. doi: 10.1002/ejp.818. Epub 2015 Oct 30. PMID 26517407
- [Background] Iannotti FA, Pagano E, Moriello AS, Alvino FG, Sorrentino NC, D'Orsi L, Gazzerro E, Capasso R, De Leonibus E, De Petrocellis L, Di Marzo V. Effects of non-euphoric plant cannabinoids on muscle quality and performance of dystrophic mdx mice. Br J Pharmacol. 2019 May;176(10):1568-1584. doi: 10.1111/bph.14460. Epub 2018 Sep 9. PMID 30074247
- [Background] Mechoulam R, Hanus L. Cannabidiol: an overview of some chemical and pharmacological aspects. Part I: chemical aspects. Chem Phys Lipids. 2002 Dec 31;121(1-2):35-43. doi: 10.1016/s0009-3084(02)00144-5. PMID 12505688
- [Background] Peres FF, Lima AC, Hallak JEC, Crippa JA, Silva RH, Abilio VC. Cannabidiol as a Promising Strategy to Treat and Prevent Movement Disorders? Front Pharmacol. 2018 May 11;9:482. doi: 10.3389/fphar.2018.00482. eCollection 2018. PMID 29867488
- [Background] Taylor L, Gidal B, Blakey G, Tayo B, Morrison G. A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Multiple Dose, and Food Effect Trial of the Safety, Tolerability and Pharmacokinetics of Highly Purified Cannabidiol in Healthy Subjects. CNS Drugs. 2018 Nov;32(11):1053-1067. doi: 10.1007/s40263-018-0578-5. PMID 30374683